CLINICAL TRIAL: NCT04066530
Title: A Randomized, Double-blinded, Active Controlled, Non-Inferiority, Multicenter, Phase III Clinical Trial to Evaluate the Efficacy and Safety of AD-203 in Patients With Acute or Chronic Gastritis
Brief Title: A Study to Evaluate the Efficacy and Safety of AD-203
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-203P3
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Acute Gastritis; Chronic Gastritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AD-203 (Experimental)
  Interventions: Drug: AD-203
- Mucosta tab. (Active Comparator)
  Interventions: Drug: Mucosta tab.

INTERVENTIONS:
Drug: AD-203 — AD-203 administered two times daily for two weeks
  Arms: AD-203
Drug: Mucosta tab. — Mucosta tab. administered three times daily for two weeks
  Arms: Mucosta tab.

SUMMARY:
This is a multicenter, active-controlled , randomized, double-blinded, paralleled group clinical study to evaluate the efficacy and safety of AD-203 to demonstrate the non-inferiority of AD-203 compared with Mucosta tab. in patients with acute or chronic gastritis

ELIGIBILITY:
Inclusion Criteria:

* Age is over 20 years old, under 75 years old, men or women
* Patients diagnosed with acute or chronic gastritis by gastroscopy

Exclusion Criteria:

* Patients who is impossible to receive gastroscopy
* Patients taking other investigational drugs or participating in other clinical studies in 3 months prior to screening visit

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
A percentage of subjects showed improvement of stomach erosions by the endoscopy. | 2 weeks
  Evaluate the improvement rate of "Very much improved' and "Much improved" of subjects with stomach erosions.
  The definition of "Very Much Improved" is the subjects showed score changed from 4 to 1 or from 3 to 1. And, "Much improved" means the subject showed score changed from 4 to 2 or from 2 to 1.

CONTACTS AND LOCATIONS:
Overall Officials: JongJae Park, Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea